CLINICAL TRIAL: NCT02832947
Title: Pharmacokinetics and Pharmacodynamics of Single Doses of Rivaroxaban in Obesity Patients Before and After Bariatric Surgery - The Extension Study
Brief Title: PK of Rivaroxaban in Bariatric Patients - Extension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 025/15_2
Record Dates: First submitted 2016-06-17; First posted 2016-07-14 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Prophylaxis of Venous Thromboembolism
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rivaroxaban Arm (Other)
  Interventions: Drug: Rivaroxaban 10 mg

INTERVENTIONS:
Drug: Rivaroxaban 10 mg — At study month 7 (+/-1 month), patients receive at 8 a.m. a single dose of 10 mg rivaroxaban. Study specific blood tubes are sampled the same day at the indicated time points from T -1h to T 12h.

SUMMARY:
Aim of this clinical Trial is the assessment of rivaroxaban PK/PD parameters in patients 6-8 months after bariatric surgery

DETAILED DESCRIPTION:
Weight loss after bariatric surgery can putatively alter drug disposition of rivaroxaban. This may be due to an altered intestinal adaptations several months after the surgical procedure. The aim of this clinical trial is to investigate pharmacokinetic and pharmacodynamic parameters after single application of 10 mg rivaroxaban in patients with prior bariatric intervention (Roux-en-y-gastric bypass or sleeve gastrectomy 6-8 months ago). PK/PD parameters will be assessed during 12 hours after application of rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Patient with past elective bariatric surgery (Roux-en-Y gastric bypass surgery or sleeve gastrectomy 6-8 months ago)
* Patient aged 18 years and older
* BMI ≥ 35 kg/m2
* Women of child-bearing age: Willingness of using a double barrier contraception method during the study
* Written, informed consent

Exclusion Criteria:

* Intake of oral anticoagulants (phenprocoumon, acenocoumarol, dabigatran, etexilate, apixaban etc.) 4 weeks prior to inclusion in the study
* Application of parenteral anticoagulants (unfractionated heparin, low molecular weight heparins, heparin derivates (fondaparinux etc.) 4 weeks prior to inclusion in the study
* Pharmacologic platelet inhibition 4 weeks prior to inclusion in the study
* Known coagulation disorders (e.g. Willebrand's disease, haemophilia)
* Evidence for deep vein thrombosis or pulmonary embolism in the personal history or in the history of first degree relatives
* Medical condition that is associated with an increased risk for VTE, i.e. active cancer disease, lupus erythematodes chronic inflammatory bowel disease
* Active, clinically significant bleeding
* Congenital or acquired bleeding disorder
* Uncontrolled severe hypertension
* Active gastrointestinal disease that can potentially lead to bleeding disorder: oesophagitis, gastritis, gastroesophageal reflux disease, chronic inflammatory bowel disease
* Vascular retinopathy
* Bronchiectasis or history of pulmonary bleeding
* Prior stroke or TIA
* Hereditary galactose intolerance, Lapp lactase deficiency, glucose-lactose malabsorption
* Severe renal impairment with a creatinine clearance (GFR) of < 30ml/min
* Positive pregnancy test, pregnancy or nursing women
* High risk of bleeding (e.g. active ulcerative gastrointestinal disease)
* Known intolerance of the study medication rivaroxaban
* Concomitant treatment with strong CYP3A4 inhibitors (e.g. ketoconazole, itraconazole, lopinavir, ritonavir, indinavir)
* Concomitant treatment with an P-glycoprotein inhibitor and weak or moderate CYP3A4 inhibitor (e.g. erythromycin, azithromycin, diltiazem, verapamil, quinidine, ranolazine, dronedarone, amiodarone, felodipine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
AUC of rivaroxaban | 1 year
Cmax of rivaroxaban | 1 year
Tmax of rivaroxaban | 1 year
Prothrombin time (PT) | 1 year
Activated partial thromboplastin time (aPTT) | 1 year
Levels of Prothrombin fragment (F1+F2) | 1 year
Levels of Thrombin-antithrombin-complexes (TAT) | 1 year
Levels of D-Dimers | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dino Kröll, MD, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital, Inselspital Berne, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No